CLINICAL TRIAL: NCT06198777
Title: Establishing Reference Intervals for Magnetocardiography Parameters in Healthy Adults in China
Brief Title: Determination of MCG Reference Intervals in Healthy Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Linyi People's Hospital (Other); Weifang People's Hospital (Other); Jining First People's Hospital (Other); Weihai Central Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); First People's Hospital of Hangzhou (Other); Chongqing Emergency Medical Center (Other); Heze Municipal Hospital (Other); Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MCG-healthy
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-12

CONDITIONS: MCG Reference Intervals Determination for Healthy Adults; Health, Subjective
Keywords: Healthy Adults; Reference Intervals

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults
  Interventions: Device: Magnetometer

INTERVENTIONS:
Device: Magnetometer — Inspection equipment for magnetocardiography

SUMMARY:
Magnetocardiography (MCG) is a promising noninvasive and accurate method for detecting cardiac abnormalities. However, the results of MCG cannot be evaluated without defined reference intervals. This is a multicenter cross-sectional study designed to establish reference values for MCG parameters healthy adults in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Those with no hospitalization for any reason in the 6 months prior to the study.
3. Those who are not currently taking any prescribed medications.
4. Those with no history of cardiovascular diseases, including coronary artery disease, structural heart disease, arrhythmia, heart failure, stroke, pulmonary embolism, aortic coarctation, or peripheral arterial disease.
5. Those with no risk factors for cardiovascular diseases, including hypertension, diabetes mellitus, hyperlipidemia.
6. Those with no history of smoking (previous non-smoking or smoking cessation >6 months).
7. Those with no excessive alcohol consumption (average daily alcohol consumption <3 drinks, 1 drink = beer 355mL / white wine 44mL / red wine 118mL).
8. Signed informed consent.

Exclusion Criteria:

1. Those with body mass index >28kg/m2 or <18kg/m2.
2. Those with resting heart rate <50 beats/min, or >110 beats/min.
3. Those with resting systolic blood pressure ≥ 140 mmHg, and/or diastolic blood pressure ≥ 90 mmHg.
4. Those with fasting blood glucose ≥7 mmol/L, and/or random blood glucose ≥11.1 mmol/L.
5. Those with total cholesterol ≥6.2 mmol/L or low-density lipoprotein cholesterol ≥4.1 mmol/L.
6. Those with abnormal electrocardiograms, such as arrhythmias, ST-T changes, and pathologic electrical axis deflections.
7. Those with cardiac ultrasonographic pathologic findings, such as left ventricular hypertrophy, left ventricular dilatation, abnormal ventricular wall motion, and valvular regurgitation or stenosis of more than mild degree.
8. Those with respiratory diseases, kidney diseases, liver diseases, endocrine diseases, anaemia or other blood diseases, connective tissue diseases, malignant tumors and other diseases.
9. Professional athletes, pregnant or lactating women, psychological or psychiatric disorders such as depression.
10. Those who are unable to perform magnetocardiography due to claustrophobia, etc., or those who are unable to cooperate with the corresponding examinations required by the study for various reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aged 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 2396 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reference value for NPM (physio-MCG parameter,%) | from the date of enrollment until the date of the completion of all assessments, up to 30 days
  MCG device is used for the measurement of the physio-MCG parameter, and we will calculate the reference value.

SECONDARY OUTCOMES:
Reference value for MCV (maximum current vector) amplitude (pT/m) at the timepoint of R wave peak | from the date of enrollment until the date of the completion of all assessments, up to 30 days
  MCG device is used for the measurement of maximum current vector amplitude (pT/m) at the timepoint of R wave peak.
Reference value for TCV (total current vector) angle at the timepoint of R wave peak | from the date of enrollment until the date of the completion of all assessments, up to 30 days
  MCG device is used for the measurement of total current vector angle at the timepoint of R wave peak.
Reference value for MCV (maximum current vector) amplitude (pT/m) at the timepoint of T wave peak | from the date of enrollment until the date of the completion of all assessments, up to 30 days
  MCG device is used for the measurement of maximum current vector amplitude (pT/m) at the timepoint of T wave peak.
Reference value for TCV (total current vector) angle at the timepoint of T wave peak | from the date of enrollment until the date of the completion of all assessments, up to 30 days
  MCG device is used for the measurement of total current vector angle at the timepoint of T wave peak.

CONTACTS AND LOCATIONS:
Overall Officials: Yuguo Chen, Professor, Principal Investigator — Qliu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China